CLINICAL TRIAL: NCT02679183
Title: Randomized Controlled Trial on Medically-Graded Honey Supplementation Formula (As a Prebiotic) To Preterm Infants
Brief Title: Medically-Graded Honey Supplementation Formula To Preterm Infants
Acronym: Honey
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem N. Said, Professor of Pediatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 100904
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Prebiotics; Honey; Premature Infants; Intestinal Microbiota
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Control 0 (Placebo Comparator): No Intervention. This group received Premature Milk Formula. This group did not receive any Medically-Graded Honey.
  Interventions: Other: Premature Milk Formula
- Group 1 (Experimental): This group received Premature Milk Formula. This group received Medically-Graded Honey (dose = 5 gram/day) for 2 weeks
  Interventions: Dietary Supplement: Medically-Graded Honey; Other: Premature Milk Formula
- Group 2 (Experimental): This group received Premature Milk Formula. This group received Medically-Graded Honey (dose = 10 gram/day) for 2 weeks
  Interventions: Dietary Supplement: Medically-Graded Honey; Other: Premature Milk Formula
- Group 3 (Experimental): This group received Premature Milk Formula. This group received Medically-Graded Honey (dose = 15 gram/day) for 2 weeks
  Interventions: Dietary Supplement: Medically-Graded Honey; Other: Premature Milk Formula

INTERVENTIONS:
Dietary Supplement: Medically-Graded Honey — Honey added to the baby formula once a day for 2 weeks.
  Arms: Group 1; Group 2; Group 3
Other: Premature Milk Formula — Enteral feeds were provided to subjects of all groups using premature milk formula as per routine nutritional management in the neonatal intensive care unit.

SUMMARY:
Honey is a natural product that contains multiple nutrients; it is composed of fructose, glucose and fructooligosaccharides that can potentially serve prebiotic functions. It also contains more than 180 substances including amino acids, vitamins, minerals and enzymes. Investigators hypothesized that supplementation of enteral feeds with honey would produce a bifidogenic effect and stimulate the immune response in preterm infants. Investigators randomly assigned subjects to 4 groups receiving 0, 5, 10 and 15 grams of honey daily for 2 weeks and measured their effect on stool colonization, systemic immune parameters and anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with gestational age ≤ 34 weeks
* postnatal age > 3 days
* no previous enteral feeding, and
* parental wish to use milk formula with no intention to use breast milk or breastfeed.

Exclusion Criteria:

* infants with major chromosomal abnormalities
* Infant with major congenital anomalies of the cardiovascular, pulmonary or central nervous system; including neuromuscular disorders and neural tube defects
* infants with intestinal atresia, tracheoesophageal fistulas, omphalocele, gastroschisis, and other major congenital GI anomalies, and
* infants with sepsis, either before or during enrollment

Ages: 3 Days to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The presence of Bifidobacterium bifidum and Lactobacillus spp in Stool | Two weeks
  Stool culture/ Gram Stain and quantitative real time PCR were used to for this outcome.

SECONDARY OUTCOMES:
CD4 and CD8 concentration in the serum | 2 weeks
  Serum concentrations of CD4 and CD8 cytokines were measured by by ELISA
Change in Weight (gram) | Baseline and 2 weeks
  The difference between weight at enrollment and at 2 weeks was measured for all subjects
Change in crown-heel length (cm) | Baseline and 2 weeks
  The difference between the length at enrollment and at 2 weeks was measured for all subjects
Change in head circumference (cm) | Baseline and 2 weeks
  The difference between head circumference at enrollment and at 2 weeks was measured for all subjects

REFERENCES:
- [Result] Boyar V, Handa D, Clemens K, Shimborske D. Clinical experience with Leptospermum honey use for treatment of hard to heal neonatal wounds: case series. J Perinatol. 2014 Feb;34(2):161-3. doi: 10.1038/jp.2013.158. PMID 24476663
- [Result] Eteraf-Oskouei T, Najafi M. Traditional and modern uses of natural honey in human diseases: a review. Iran J Basic Med Sci. 2013 Jun;16(6):731-42. PMID 23997898
- [Result] Ezz El-Arab AM, Girgis SM, Hegazy EM, Abd El-Khalek AB. Effect of dietary honey on intestinal microflora and toxicity of mycotoxins in mice. BMC Complement Altern Med. 2006 Mar 14;6:6. doi: 10.1186/1472-6882-6-6. PMID 16533410
- [Result] Kapiki A, Costalos C, Oikonomidou C, Triantafyllidou A, Loukatou E, Pertrohilou V. The effect of a fructo-oligosaccharide supplemented formula on gut flora of preterm infants. Early Hum Dev. 2007 May;83(5):335-9. doi: 10.1016/j.earlhumdev.2006.07.003. Epub 2006 Sep 14. PMID 16978805
- [Derived] Aly H, Said RN, Wali IE, Elwakkad A, Soliman Y, Awad AR, Shawky MA, Alam MSA, Mohamed MA. Medically Graded Honey Supplementation Formula to Preterm Infants as a Prebiotic: A Randomized Controlled Trial. J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):966-970. doi: 10.1097/MPG.0000000000001597. PMID 28379925